CLINICAL TRIAL: NCT06173492
Title: The Use of Platelet-Rich Fibrin as Solely Filling Material in Socket Preservation Technique: a Randomized-controlled Clinical Trial
Brief Title: Platelet Rich Fibrin (PRF) in Socket Preservation Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Naples (Other)
Responsible Party: Principal Investigator, Gilberto Sammartino, Full professor, University of Naples
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNaples 401-19
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Alveolar Bone Loss; Tooth Extraction
Keywords: Dental implant; Socket ridge preservation; Platelet Rich Fibrin
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Tooth Extraction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Socket ridge preservation with PRF (Experimental): 40 ml of blood is drawn and collected in plastic tubes of 10 ml. The tubes are placed in a centrifuge at 2700 rpm for 12 minutes to get the clot of fibrin. After extraction, the clot obtained by centrifugation is made into PRF cylinders and inserted into the socket and compacted.
  Interventions: Procedure: Dental extraction; Device: Platelet Rich Fibrin
- Spontaneous healing (Active Comparator): No treatment is applied. The socket is made to heal spontaneously.
  Interventions: Procedure: Dental extraction

INTERVENTIONS:
Procedure: Dental extraction — After local anesthesia (mepivacaine 2%), the tooth is extracted atraumatically with levers and forceps taking care to preserve the cortex. The roots of multi-rooted teeth are separated before extraction. The pocket epithelium and granulation tissue inside the socket are removed.
Device: Platelet Rich Fibrin — The clot obtained by centrifugation is made into PRF cylinders and inserted into the socket and compacted.
  Arms: Socket ridge preservation with PRF

SUMMARY:
The loss of a tooth or change in its function is lead to a change in alveolar ridge's height and volume. Socket preservation (SP) is a procedure designed to prevent or limit alteration of the post-extraction bone ridge to achieve an optimal prosthetic implant rehabilitation. The aim of this randomized-controlled clinical trial is to suggest that platelet rich fibrin (PRF) as solely grafting material may be a valid tool in this technique.

DETAILED DESCRIPTION:
80 patients with mandibular or maxillary premolars that need to be extracted will be recruited. All patients will be randomly treated by using two different therapeutic approaches, thereby yielding two different study groups, each of which is composed of 40 cases: in the test group the socket preservation technique with PRF will be performed, in control group the post-extraction socket is left healing spontaneously without performing socket preservation.

A software will be used to produce a random sequence of 80 integer numbers without duplicates generated by a software and concealed in closed envelopes by one of the investigators. At the time of the patient's first surgery, the envelope will be opened and patient allocated either to test or control group. All patients are informed by the written consent obtained that they could be causally allocated to one of the two groups.

Before extraction, patients should undergo to periodontal treatment and instrumental investigations such as orthopantomography.

After local anesthesia (mepivacaine 2%), the tooth is extracted atraumatically with levers and forceps taking care to preserve the bone cortex. The roots of multi-rooted teeth are separated before extraction. The pocket epithelium and the granulation tissue are removed.

In the test group, a blood collection of 40 ml will be performed and PRF is made according to the manufacturer instructions.

One clinician, not involved in patient treatment and not aware of what therapeutic approach used for the different sites of treatment, will perform all clinical measurements immediately after surgery and three months later.

Patients will be checked at 3 days, 1 week after surgery (removal of sutures), 14 days after surgery, 28 days after surgery and at 3 months after surgery (at the time of implant placement).

A Cone Beam Computed Tomography (CBCT) is prescribed immediately after surgery and 3 months after surgery before implant placement.

Differences between the two analysed groups will be evaluate by test t-student through a statistic software.

ELIGIBILITY:
Inclusion Criteria:

* Mandibular or maxillary premolars that need to be extracted due to endodontic failure, caries or fractures and will need to be replaced with a dental implant after 3 months of healing
* Full mouth plaque score ≤ 25% at onset
* Full mouth bleeding score ≤ 25% at onset
* Integrity of the alveolar walls after extraction
* Vestibular wall thickness < 1 mm
* Patients able to understand and sign informed consensus

Exclusion Criteria:

* Significant medical conditions contraindicating surgery
* Pregnancy and breastfeeding
* Tobacco smoking (>15 cigarettes per day)
* Immunocompromised patients
* Alcohol and drug abuse
* Uncooperative patients
* Periodontally compromised patients
* Acute abscesses at the extraction site
* Other dental elements that are not premolars
* Patients who do not show up for scheduled checkups

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Periodontal probe - alveolar crest distance | Immediately after surgery, 3 months after surgery
  Vertical distance measured with a periodontal probe from the alveolar crest (AC) to a reference periodontal probe (P) connecting the cement-enamel junction (CEJ) of the teeth adjacent.
Width | Immediately after surgery, 3 months after surgery
  Horizontal alveolar ridge thickness from the external face of the buccal wall to the outer face of the lingual side is measured with a hand caliper, 1 mm apically from the alveolar ridge in the central area.
Vestibular bone wall thickness | Immediately after surgery, 3 months after surgery
  It is measured with a hand caliper at the center of the vestibular wall, 1 mm apically from the ridge.

SECONDARY OUTCOMES:
Wound healing index | 3, 7, 14, 28 days after surgery
  Landry index including description from a "Very poor" to an "Excellent" wound healing

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto Sammartino, Principal Investigator — Federico II University
Locations (1):
- Gilberto Sammartino, Naples, Italy

REFERENCES:
- [Result] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Result] Chiapasco M, Zaniboni M, Rimondini L. Dental implants placed in grafted maxillary sinuses: a retrospective analysis of clinical outcome according to the initial clinical situation and a proposal of defect classification. Clin Oral Implants Res. 2008 Apr;19(4):416-28. doi: 10.1111/j.1600-0501.2007.01489.x. Epub 2008 Feb 11. PMID 18266875
- [Result] Dohan Ehrenfest DM, de Peppo GM, Doglioli P, Sammartino G. Slow release of growth factors and thrombospondin-1 in Choukroun's platelet-rich fibrin (PRF): a gold standard to achieve for all surgical platelet concentrates technologies. Growth Factors. 2009 Feb;27(1):63-9. doi: 10.1080/08977190802636713. PMID 19089687
- [Result] Cortellini P, Pini Prato G, Baldi C, Clauser C. Guided tissue regeneration with different materials. Int J Periodontics Restorative Dent. 1990;10(2):136-51. No abstract available. PMID 2084057
- [Result] Zhang Y, Ruan Z, Shen M, Tan L, Huang W, Wang L, Huang Y. Clinical effect of platelet-rich fibrin on the preservation of the alveolar ridge following tooth extraction. Exp Ther Med. 2018 Mar;15(3):2277-2286. doi: 10.3892/etm.2018.5696. Epub 2018 Jan 4. PMID 29456635
- [Result] Maiorana C, Poli PP, Deflorian M, Testori T, Mandelli F, Nagursky H, Vinci R. Alveolar socket preservation with demineralised bovine bone mineral and a collagen matrix. J Periodontal Implant Sci. 2017 Aug;47(4):194-210. doi: 10.5051/jpis.2017.47.4.194. Epub 2017 Aug 11. PMID 28861284